CLINICAL TRIAL: NCT02732301
Title: Gastrointestinal Dysfunktion Efter hjärtkirurgi - förekomst Samt sökande Efter Nya biomarkörer
Brief Title: Postoperative Gastrointestinal Dysfunction After Cardiac Surgery - Occurrence and Search for Biomarkers
Acronym: GAINDYSFUNCS
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Region Örebro County (Other)
Responsible Party: Sponsor
Other Study IDs: 188051
Record Dates: First submitted 2016-04-04; First posted 2016-04-08 (Estimated); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Thoracic Surgical Procedures; Gastrointestinal Tract; Cardiopulmonary Bypass; Biomarkers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Four plasma samples, 2 ml each, taken preoperatively and the three first postoperative days, which are stored in an approved biobank.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to investigate the frequency and grade of gastrointestinal dysfunction in patients after thoracic cardiovascular surgery, and to search for biomarkers of gastrointestinal dysfunction. All adult patients undergoing elective cardiac surgery requiring cardiopulmonary bypass at Örebro University Hospital, Örebro, Sweden, are asked for participation in this study. All participating patients sign informed consent at the inclusion. The first three postoperative days the function of the gastrointestinal tract is scored according to a rating scale (grade 0-4), along with other clinical parameters. Plasma blood samples are collected from each patient preoperatively and the first three postoperative days. The plasma samples are stored in a biobank for later determination of plasma proteins. In the analysis, the patients are divided according to the gastrointestinal rating scale and the plasma protein expression, gastrointestinal complications and all-cause mortality are compared between the groups.

ELIGIBILITY:
Inclusion Criteria:

* Accepted for an elective thoracic cardiovascular surgical procedure requiring cardiopulmonary bypass
* >18 years old

Exclusion Criteria:

* Present and severe symptoms from the gastrointestinal tract
* Previous major/extensive abdominal surgery
* Presence of astomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing elective thoracic cardiovascular surgical procedures requiring intraoperative cardiopulmonary bypass at Örebro University Hospital, Örebro, Sweden, using a consecutive sampling method.
Sampling Method: Probability Sample
Enrollment: 501 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Acute gastrointestinal injury score | Postoperative days 1-3
  Acute gastrointestinal injury score from Reintam Blaser et al (2012) modified for postoperative patients.

SECONDARY OUTCOMES:
Plasma protein expression | Postoperative days 1-3
Gastrointestinal complications | 30 days postoperative
All cause mortality | 30 days postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Kristofer F Nilsson, MD, PhD, Principal Investigator — Department of Cardio-Thoracic and Vascular Surgery, Örebro University Hospital, Örebro, SWEDEN
Locations (1):
- Department of Cardio-Thoracic and Vascular Surgery, Örebro University Hospital, Örebro, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Reintam Blaser A, Malbrain ML, Starkopf J, Fruhwald S, Jakob SM, De Waele J, Braun JP, Poeze M, Spies C. Gastrointestinal function in intensive care patients: terminology, definitions and management. Recommendations of the ESICM Working Group on Abdominal Problems. Intensive Care Med. 2012 Mar;38(3):384-94. doi: 10.1007/s00134-011-2459-y. Epub 2012 Feb 7. PMID 22310869